CLINICAL TRIAL: NCT04273503
Title: Healthy Immigrant Community: Pilot Social Network Weight Loss Intervention
Brief Title: Pilot Social Network Weight Loss Intervention
Acronym: HIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark L Wieland, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-011574
Record Dates: First submitted 2020-02-12; First posted 2020-02-18 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Diet, Healthy; Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Behavioral intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will receive education on maintaining a healthy diet and improving physical activity.
  Interventions: Behavioral: Mentoring/educational session

INTERVENTIONS:
Behavioral: Mentoring/educational session — 12 mentoring/educational sessions focused on physical activity and healthy nutrition by Mayo Clinic experts.

SUMMARY:
Specific Aim #1: Pilot test a social network-informed CBPR-derived health promotion program for feasibility outcomes with overweight or obese adults from two immigrant communities.

Specific Aim #2: Assess the preliminary impact of embedding a social network-informed CBPR-derived intervention within a regional health promotion resource hub on sustainability and uptake outcomes.

DETAILED DESCRIPTION:
The intervention will consist of 12 community-based mentoring and education sessions, group activities and application of a community toolkit for healthy weight loss delivered by trained interventionists from Hispanic and Somali communities to their social networks. Using a pre-post study design, 4 social networks of adults with approximately 32 network participants will receive the intervention. Primary outcomes, measured 3 months after implementation, will include feasibility measures of acceptability, implementation, and practicality. Secondary outcomes will include BMI, waist circumference, blood pressure, fasting blood glucose, total cholesterol, physical activity level, dietary change, and health-related quality of life.

Eligibility criteria include (1) self-identification as Hispanic or Somali, (2) member of an HPs social network, (3) age≥18 and <65 (4) willingness to participate in all aspects of the study; and (5) provision of informed consent. Exclusion criteria include (1) pregnancy at the time of enrollment and (2) serious medical conditions or disabilities that would make physical activity difficult.

We will test how best to integrate a social network intervention within an existing evidence-based regional health promotion infrastructure (WellConnect) that will enhance its potential dissemination and community-wide uptake

ELIGIBILITY:
Inclusion Criteria:

1. self-identification as Hispanic or Somali
2. member of an HPs social network
3. age≥18 and <65
4. willingness to participate in all aspects of the study
5. provision of informed consent.

Exclusion Criteria:

1. pregnancy at the time of enrollment
2. serious medical conditions or disabilities that would make physical activity difficult.

   * To avoid stigmatization, a normal weight (BMI<25) will not exclude individuals from participating, but they will be excluded from the measurements and analyses.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability | 12 weeks
  To what extent did was the intervention judged as relevant, satisfying, or helpful to HPs and participants? Interviews with HPs; focus groups and survey with participants.

SECONDARY OUTCOMES:
Weight | 12 weeks
  Weight will be measured to the nearest 0.1 kg using a portable scale (Seca 880 Digital Floor Scale). BMI is calculated as weight (kg)/height squared (m2).
Waist circumference | 12 weeks
  Waist circumference will be measured to the nearest 0.1 cm at the narrowest part of the torso between the ribs and the iliac crest. Participants will remove all excess clothing prior to the measurement and smooth the remaining clothing against the skin. Two measurements will be taken; if the difference between the two measures is more than 2.0 cm, a third measurement will be taken. The average of the two closest measures will be used for analyses.
Glucose | 12 weeks
  Collected by a single finger prick. Participants will be asked to refrain from eating for at least 6 hours prior to testing. Samples used for testing are whole blood from a fingerstick collected in a lithium heparin coated capillary tube.
Cholesterol | 12 weeks
  Collected by a single finger prick. Participants will be asked to refrain from eating for at least 6 hours prior to testing. The portable Whole Blood Lipid Screen Cholestech LDX Analyzer will be used to analyze specimens, which combines enzymatic methodology and solid-phase technology measured by reflectance photometry to measure total cholesterol, HDL cholesterol, triglycerides and glucose in whole blood. LDL cholesterol is a calculated value. Samples used for testing are whole blood from a fingerstick collected in a lithium heparin coated capillary tube. Results will be recorded at the site of collection and samples will be destroyed upon recording of results.
Height | 12 weeks
  Height will be measured to the nearest 0.1 cm at baseline only using a stadiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wieland, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials